CLINICAL TRIAL: NCT06642038
Title: Efficacy and Safety of Transbronchial BTVA in Heterogeneous Emphysema: A Prospective, Single-Arm, Multicenter Clinical Study
Brief Title: Efficacy and Safety of Transbronchial Bronchoscopic Thermal Vapor Ablation (BTVA) in Heterogeneous Emphysema
Status: Not yet recruiting | Type: Observational
Sponsor: Ye Gu (Other)
Collaborators: Ruijin Hospital (Other); First Hospital of China Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Shandong Provincial Public Health Clinical Center (Unknown); First Affiliated Hospital, Sun Yat-Sen University (Other); Zhongda Hospital (Other); Jiangxi Provincial People's Hopital (Other); Shenzhen Baoan District People 's Hospital (Unknown); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor-Investigator, Ye Gu, Principal Investigator, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Other Study IDs: L23-399
Record Dates: First submitted 2024-09-29; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Heterogeneous Emphysema
Keywords: BTVA; Heterogeneous emphysema; Bronchoscopy; Efficacy and Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental Group
  Interventions: Procedure: Transbronchial Endoscopic Thermal Vapor Ablation

INTERVENTIONS:
Procedure: Transbronchial Endoscopic Thermal Vapor Ablation — Transbronchial Endoscopic Thermal Vapor Ablation

SUMMARY:
Efficacy and Safety of Transbronchial BTVA in Heterogeneous Emphysema: A Prospective, Single-Arm, Multicenter Clinical Study

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥40 and ≤75 years old
2. Heterogeneous emphysema
3. 20% predicted value ≤ FEV1 ≤ 50% predicted value, TLC ≥ 100% predicted value, RV ≥ 150% predicted value, DLCO ≥ 20% predicted value
4. 6-minute walking distance (6MWD) > 140m
5. mMRC index ≥ 2
6. The patients have fully understood the content of the trial and voluntarily signed the informed consent form

Exclusion Criteria:

1. Contraindications to bronchoscopy include: myocardial infarction within the past month, active massive hemoptysis, coagulation dysfunction, pregnancy, malignant arrhythmia, severe pulmonary hypertension, extreme systemic failure, and other conditions
2. Concomitant diseases that may significantly increase the risk of complications after BTVA treatment include, but are not limited to: immune system disorders, bleeding disorders, unstable cardiovascular disease, a history of asthma, and alpha-1 antitrypsin deficiency
3. Concomitant medications known to significantly increase the risk of complications after BTVA treatment include, but are not limited to: immunosuppressive drugs (except topical medications), anticoagulants, and antiplatelet drugs
4. Receiving morphine derivatives within 4 weeks prior to screening
5. Respiratory tract infection or exacerbation of chronic obstructive pulmonary disease (COPD) within 6 weeks prior to screening
6. The upper and lower lobes of the other lung have high-grade emphysematous lesions, defined as HRCT showing that the low-density attenuation area (less than -950 Hu) accounts for more than 40% of the total lung volume.
7. The lobe of the lung where the intended treatment segment is located has large bullae (defined as bullae that occupy more than one-third of the lobe) or paralobular septal emphysema.
8. Symptoms or abnormal laboratory values suggesting active infection (e.g., fever, elevated white blood cell count, etc.).
9. Patients who have undergone or plan to undergo lung or chest surgery during this study, including but not limited to lung resection or lung transplantation.
10. Patients evaluated by specialists to have highly suspected malignant pulmonary nodules.
11. Women who intend to become pregnant, are pregnant, or are breastfeeding during the study.
12. Patients participating in other drug or medical device clinical trials.
13. The investigator believes the patient has other conditions that make them unsuitable for inclusion in this study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are planning to receive BTVA for heterogeneous emphysema
Sampling Method: Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2024-10-13 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The forced expiratory volume in one second (FEV1) is used to assess lung function | 6 months
  Evaluate the improvement in FEV1 from baseline to 6 months after BTVA treatment.
The Saint George's Respiratory Questionnaire-C (SGRQ-C) questionnaire was used to evaluate the value of patients' quality of life. | 6 months
  Evaluate the improvement in SGRQ-C questionnaire from baseline to 6 months after BTVA treatment. The total score of SGRQ-C questionnaire usually ranges from 0 to 100, with 0 representing the best condition and 100 representing the worst condition.

SECONDARY OUTCOMES:
FEV1 is used to assess lung function | 12 months
  Improvement in FEV1 12 months after the first treatment.
The SGRQ-C questionnaire was used to evaluate the value of patients' quality of life. | 12 months
  Improvement in SGRQ-C 12 months after the first treatment. The total score of SGRQ-C questionnaire usually ranges from 0 to 100, with 0 representing the best condition and 100 representing the worst condition.
Forced expiratory volume in one second/Forced vital capcacity（FEV1/FVC） were used to assess lung function | 6 and 12 months
  Improvement in FEV1/FVC compared to baseline at 6 and 12 months after the first treatment
FVC were used to assess lung function | 6 and 12 months
  Improvement in FVC compared to baseline at 6 and 12 months after the first treatment
ResidualVolume (RV) were used to assess lung function | 6 and 12 months
  Improvement in RV compared to baseline at 6 and 12 months after the first treatment
Total Lung Capacity（TLC） were used to assess lung function | 6 and 12 months
  Improvement in TLC compared to baseline at 6 and 12 months after the first treatment
6 minute walking distance (6MWD) was used to assess exercise tolerance | 6 and 12 months
  Improvement in exercise tolerance compared to baseline at 6 and 12 months after the first treatment: 6MWD.
Symptom scoring using COPD Assessment Test (CAT), modified Medical Research Council （mMRC） scoring table | 6 and 12 months
  Improvement in symptom scores compared to baseline at 6 and 12 months after the first treatment: CAT, mMRC. The CAT score is a comprehensive assessment of symptoms, ranging from 0 to 40 points. A score of 10 or above indicates a higher number of symptoms. Scores between 0 and 10 reflect a mild impact, 11 to 20 indicate a moderate impact, 21 to 30 represent a severe impact, and 31 to 40 signify a very severe impact on the patient's condition. The mMRC score is a scale used to assess the degree of breathlessness, with a range from 0 to 4. A higher score indicates greater severity of symptoms. A score of 0 reflects no breathlessness except with strenuous exercise, 1 indicates breathlessness when hurrying on level ground or walking up a slight hill, 2 represents breathlessness causing the patient to walk slower than people of the same age or having to stop for breath when walking at their own pace, 3 indicates stopping for breath after walking about 100 meters or after a few minutes on le
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | At surgery and 12 months after surgery
  All adverse events during surgery and postoperative follow-up were recorded and evaluated according to CTCAE V5.0. The relevance of these events to BTVA treatment was assessed, and the incidence of adverse events and serious adverse events related to BTVA treatment was calculated.

IPD SHARING:
Plan to Share IPD: No
The dataset produced during this study is available upon request from the corresponding author (drsymons@outlook.com).